CLINICAL TRIAL: NCT06144710
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Characteristics of SG301 SC Injection in Single-dose Healthy Subjects and Multiple-dose Systemic Lupus Erythematosus (SLE) Subjects
Brief Title: SG301-SC Injection Safety Study in Subjects With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSG-301 SC-101
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: This Study consists of Parts A and B. Part A ：Single dose of SG301 SC Injection in healthy volunteers. This part will consist of 1 mg/kg dose group (n=4) and 2 mg/kg dose group(n=4) , all 4 participants in each group will receive a single dose of SG301 SC Injection by abdominal subcutaneous injection.
  Part B：Multiple doses of SG301 SC Injection/SG301 SC placebo in SLE patients. The MAD will be performed at a ratio of 8:2 in 4 dose groups (n=10/group), namely 2 mg/kg, 4 mg/kg, 8 mg/kg, and 12 mg/kg dose groups. The SG301 SC Injection or SG301 SC placebo will be subcutaneously injected every 2 weeks [Q2W] in a 2-week cycle for a total of 6 doses in the MAD study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part A：Open-label Part B：Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SG301 SC (Experimental): Part A: Dose escalation of SG301 SC will be done in healthy volunteers at 1 mg/kg dose group and 2 mg/kg dose group.
  Part B: Dose escalation of SG301 SC will be done in Systemic lupus erythematosus subjects in 4 dose groups, namely 2 mg/kg, 4 mg/kg, 8 mg/kg, and 12 mg/kg dose groups. 8 subjects will be randomized to SG301 SC injection in an 8:2 ratio at each dose group.
  Interventions: Drug: SG301 SC Injection
- Placebo (Placebo Comparator): Part B: Dose escalation of SG301 SC will be done in Systemic lupus erythematosus subjects in 4 dose groups, namely 2 mg/kg, 4 mg/kg, 8 mg/kg, and 12 mg/kg dose groups. 2 subjects will be randomized to SG301 SC injection in an 8:2 ratio at each dose group.
  Interventions: Drug: SG301 SC Injection; Drug: SG301 SC Placebo

INTERVENTIONS:
Drug: SG301 SC Injection — Subcutaneous injection every two weeks
Drug: SG301 SC Placebo — Subcutaneous injection every two weeks
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I clinical study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single dose in healthy volunteers and multiple doses of SG301 SC injection in participants with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a phase I single ascending dose (SAD) study in healthy volunteers and multiple ascending dose (MAD) study in participants with mild or moderate SLE, which consists of Parts A and B. Part A adopts a single-center, open-label, dose escalation trial design, and Part B adopts a multi-center, randomized, double-blind, placebo-controlled trial design to evaluate the safety, tolerability, PK, and immunogenicity, preliminary efficacy of SG301 SC Injection in patients with mild to moderate SLE.

ELIGIBILITY:
Inclusion Criteria:

Part A (healthy volunteers)

1. Male healthy adults aged 18-50 years (inclusive);
2. Male participants weighed 50-100 kg (inclusive) with the body mass index of 19.0-27.0 kg/m2 (inclusive);
3. Participants whose partners are of childbearing potential must agree to use effective contraceptive methods throughout the study period and for 6 months following the last dose.

Part B (SLE participants)

1. Males or females aged 18-65 years (inclusive);
2. BMI 18.5-30.0 kg/m2 (inclusive);
3. Have diagnosed as SLE based on the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) SLE classification criteria, with inadequate response or intolerance to or having relapsed despite the standard treatment;
4. SELENA-SLEDAI score >4 and ≤12;
5. Serologically ANA and/or anti-ds-DNA antibody tested positive;
6. Having received a standard treatment for at least 12 weeks prior to the first dose that has remained at a stable dose for at least 4 weeks prior to the first dose;
7. Laboratory values at screening meets the following criteria:

   1. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2ULN, total bilirubin <1.5×ULN;
   2. Renal function: creatinine (Cr) and urea ≤1.5×ULN; eGFR >60 ml/min (calculated by the MDRD formula); urine total protein-creatinine ratio ≤3.0 g/g or 24h urine protein ≤3.5 g;
   3. Bone marrow function: Hb≥100g/L, WBC≥3.0×109/L, PLT≥75×109/L;
   4. Participants who are of childbearing potential or whose partners are of childbearing potential must agree to use effective contraceptive methods throughout the study period and for 6 months following the last dose.

Exclusion Criteria:

Part A (healthy volunteers)

1. Have a history of allergies or likely to be allergic to the investigational drug or any of their ingredients judged by the investigators;
2. Have previously received drugs of the same target (CD38);
3. Have participated in a clinical trial of any drug or medical device within 3 months or 5 half-lives prior to dosing, whichever is longer;
4. Have received any prescription drugs or Chinese herbal medicines within 4 weeks prior to dosing, or any non-prescription or dietary supplements within 2 weeks prior to dosing;
5. Have infections within 2 weeks prior to first dose (including but not limited to viral, bacterial, or fungal infections);
6. Have experienced symptomatic herpes zoster within 3 months prior to dosing;
7. Presence of any of the following diseases assessed by the investigator as abnormal with clinical significance within 6 months prior to dosing;
8. Have a history of cardiovascular diseases within 6 months prior to dosing: chronic congestive heart failure (New York Heart Association [NYHA] Class III or IV), myocardial infarction, severe heart diseases (e.g., unstable angina, cardiogenic shock, arrhythmias requiring treatment, heart valve diseases, hypertrophic cardiomyopathy, and rheumatic heart disease, etc.), and familial long QT interval syndrome, etc.;
9. Presence of chronic nervous system symptoms such as dizziness and headache prior to dosing;
10. Blood cell count below the lower limit of normal (LLN), or clinically significant abnormalities in any other hematology tests within 1 week prior to dosing;
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.2×ULN, total bilirubin >1.2×ULN;
12. ECG abnormalities with clinical significance, e.g. QTcF >450 ms;
13. Any vital signs abnormal with clinical significance;
14. Fasting blood glucose above ULN;
15. Any abnormal from physical examination, laboratory tests, or chest CT with clinical significance;
16. Hepatitis B surface antigen (HBsAg) or core antibody (HBcAb) positive, hepatitis C virus (HCV) antibody positive, TPPA positive, or HIV antibody positive;
17. Mycobacterium tuberculosis infection;
18. Having received a live or attenuated live vaccine within 4 weeks prior to dosing or planning to do so during the trial;
19. Skin injection site abnormal, including but not limited to birthmarks, scars, black moles, tattoos, and open wounds;
20. Blood donation ≥400 ml or blood loss ≥400 ml within 4 weeks prior to dosing, or having received blood transfusion within 8 weeks prior to dosing;
21. A history of heavy drinking within 3 months prior to dosing;
22. A history of drug abuse within 5 years prior to dosing or use of narcotics within 3 months prior to the trial.

Part B (SLE participants)

1. Has a history of central nervous system disorders that require prohibited medicine treatment within 2 months prior to the first dose;
2. Presence of concomitant rheumatic diseases within 12 months prior to the first dose, including but not limited to rheumatoid arthritis, spondyloarthritis, dermatomyositis/polymyositis, Sjogren's syndrome, systemic sclerosis, mixed connective tissue disease, and overlap syndrome, etc.;
3. Presence of catastrophic antiphospholipid syndrome within 12 months prior to the first dose;
4. Has a history of non-SLE inflammatory skin or joint disease within 12 months prior to the first dose;
5. Presence of chronic active infection or acute infection within 4 weeks prior to first dose or superficial skin infection within 1 week prior to first dose;
6. A known or suspected history of immunosuppression;
7. Have undergone a major surgery within 12 weeks prior to the first dose or having an unhealed wound, ulcer or fracture, or planning to undergo a major surgery during the study;
8. Having participated in any clinical trial within 12 weeks prior to the first dose or have received other investigational products within 5 half-live, whichever is longer;
9. Have received any drugs targeting T or B lymphocytes (e.g., rituximab) within 6 months or cytokines or cytokines receptors (e.g., belimumab, telitacicept, etc.) treatment within 5 half-lives prior to the first dose;
10. Having received JAK inhibitors treatment within 12 weeks or 5 half-lives prior to the first dose, whichever is shorter;
11. Having received any of the following treatment within 12 weeks prior to the first dose:

    1. Intravenous immunoglobulin (IVIG)
    2. Plasma exchange
    3. Intravenous cyclophosphamide;
12. Have diseases with major clinical significance within 6 months prior to first dose, including but not limited to circulatory system disorders, endocrine system disorders, nervous system disorders, blood system disorders, immune system disorders, and psychiatric disorders, etc.;
13. A history of cardiovascular diseases within 6 months prior to the first dose, including but not limited to chronic congestive heart failure (NYHA Class III or IV), myocardial infarction, severe heart diseases (e.g., unstable angina, cardiogenic shock, arrhythmias requiring treatment, heart valve diseases, hypertrophic cardiomyopathy, and rheumatic heart disease, etc.), QTcF >450 ms or familial long QT interval syndrome, poorly controlled hypertension;
14. Mycobacterium tuberculosis infection;
15. Presence of active hepatitis:

    1. HBsAg positive and/or HBcAb positive and HBV DNA positive;
    2. HCV antibody positive and HCV RNA positive;
16. HIV antibody positive;
17. Both TPPA and RPR positive;
18. Known allergy to monoclonal antibody drugs or to any excipient of the investigational drug;
19. Having received a live or attenuated live vaccine within 4 weeks prior to the first dose or planning to do so during the study;
20. Have a history of major organ transplantation or hematopoietic stem cell/ bone marrow transplantation;
21. Have a history of malignancy within 5 years prior to first dose;
22. Participants with depression or suicidal tendency;
23. Have a history of heavy drinking or drug abuse within 3 months prior to first dose;
24. Pregnant or breastfeeding women, or women who plan to become pregnant or may breastfeed during the study and for 6 months following the last dose; male participants whose partner plans to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events(Part A and Part B) | From baseline through the end of study. Part A: Average 2 months per subject, Part B: Average 5 months per subject.
  Number and percentage of AEs which are calculated by worst CTCAE grade by CTCAE 5.

SECONDARY OUTCOMES:
RP2D (PartB) | From baseline through the end of study. Average 5 months per subject.
  RP2D will be determined based on the DLTs and safety data.
Pharmacokinetics (PK): Cmax (Part A and Part B) | From baseline through the end of study. Part A: Average 2 months per subject, Part B: Average 5 months per subject.
  Cmax to maximum drug concentration administration.
Pharmacokinetics (PK): limination half-life (T1/2) (Part A and Part B) | From baseline through the end of study. Part A: Average 2 months per subject, Part B: Average 5 months per subject.
  Limination half-life (T1/2) of the drug after administration.
Immunogenicity (Part A and Part B) | From baseline through the end of study. Part A: Average 2 months per subject, Part B: Average 5 months per subject.
  Anti-SG301 antibody (ADAdrug), neutralizing antibody (Nabdrug, to be detected only in case of the presence of ADAdrug), and anti-hyaluronidase antibody (ADArHu).
PD endpoints: CD38 RO (Part B) | From baseline through the end of study. Average 5 months per subject.
  Detect the CD38 RO
Biomarkers evaluation (Part B) | From baseline through the end of study. Average 5 months per subject.
  It includes anti-ds-DNA autoantibody and complement factors C3 and C4.
Efficacy evaluation (Part B) | From baseline through the end of study. Average 5 months per subject.
  Activity will be evaluated by SELENA SLEDAI.
Evaluation of exploratory measures：immunoglobulins (Part B) | From baseline through the end of study. Average 5 months per subject.
  Changes from baseline in immunoglobulins IgG, IgM and IgA with the investigational drug SG301 SC Injection and SG301 SC placebo.
Evaluation of exploratory measures：BILAG-2004 /PGA (Part B) | From baseline through the end of study. Average 5 months per subject.
  Changes from baseline in BILAG-2004 and PGA with the investigational drug SG301 SC Injection and SG301 SC placebo.
Evaluation of exploratory measures：immune cell (Part B) | From baseline through the end of study. Average 5 months per subject.
  Changes from baseline in the immune cell subsets including NK cells (activated and total), B cell subsets, plasmacytes, and plasmablasts, etc.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No